CLINICAL TRIAL: NCT00511940
Title: Acamprosate in the Treatment of Binge-Eating Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Forest Laboratories (Industry); University of Cincinnati (Other)
Responsible Party: Susan L. McElroy, MD, Lindner Center of HOPE
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMP-MD-20
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): acamprosate
  Interventions: Drug: acamprosate
- 2 (Placebo Comparator): sugar pill
  Interventions: Other: placebo

INTERVENTIONS:
Drug: acamprosate — 999 mg/day - 2997 mg/day, oral
  Other Names: Campral
  Arms: 1
Other: placebo — oral, placebo
  Arms: 2

SUMMARY:
The purpose of this research study is to determine the efficacy (how well it works), tolerability and safety of acomprosate compared with placebo in patients with binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet the DSM-IV (1) criteria for a diagnosis of binge eating disorder (BED) for at least the last 6 months. The DSM-IV criteria are as follows:

  * Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following: eating, in a discrete period of time (eg, within any two hour period), an amount of food that is definitely larger than most people would eat in a similar period of time under similar conditions; and a sense of lack of control over eating during the episode (eg, a feeling that one cannot stop eating or control what or how much one is eating).
  * The binge eating episodes are associated with at least three of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.
  * Marked distress regarding binge eating.
  * The binge eating occurs, on average, at least two days a week for six months.
  * The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
* In addition, subjects will report at least 3 binge eating episodes per week for the last 6 months prior to randomization
* Weight > 85% of the midpoint of ideal body weight for their height. (According to the Metropolitan Height/Weight table.) The subject population is expected to include both normal weight and obese individuals (although the majority of subjects are expected to be overweight).
* Men or women, between the ages of 18 and 65. The subject population is expected to be predominantly made up of women.

Exclusion Criteria:

* Have concurrent symptoms of bulimia nervosa or anorexia nervosa, including weight loss to at least 15% below the Metropolitan Height/Weight tables.
* Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. (All women of childbearing potential will have a negative pregnancy test before entering the study).
* Patients who are displaying clinically significant suicidality or homicidality.
* Patients who have received psychotherapy or behavioral therapy from a mental health professional as a part of previous treatment for BED for at least 3 months prior to randomization.
* A DSM-IV diagnosis of substance abuse or dependence (except nicotine abuse or dependence) within the 6 months prior to randomization.
* A lifetime DSM-IV history of psychosis, mania or hypomania, or dementia.
* History of any psychiatric and personality disorder (eg, schizotypal and borderline) which might interfere with a diagnostic assessment, treatment, or compliance.
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease which could interfere with diagnosis, treatment, or assessment of BED. Patients should be biochemically euthyroid to enter the study.
* History of seizures, including febrile seizures in childhood.
* Patients requiring treatment with any drug which might interact adversely with or obscure the action of the study medication.
* Clinically relevant abnormal laboratory results, specifically including hypokalemia.
* Patients who have received monoamine oxidase inhibitors, antipsychotics, lithium, or fluoxetine within four weeks prior to randomization.
* Patients who have received other psychoactive medications (other than hypnotics) within one week prior to randomization.
* Patients who have received investigational medications or depot neuroleptics within three months prior to randomization.
* Patients previously enrolled in this study or have previously been treated with acamprosate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be change in weekly binge frequency | 10 weeks

SECONDARY OUTCOMES:
Secondary efficacy variables will include change in binge day frequency (days during which at least one binge occurs), obsessive-compulsive symptoms of BED, craving for food, depressive symptoms, weight, and BMI | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McElroy, MD, Principal Investigator — Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Guerdjikova AI, Winstanley EL, O'Melia AM, Mori N, McCoy J, Keck PE Jr, Hudson JI. Acamprosate in the treatment of binge eating disorder: a placebo-controlled trial. Int J Eat Disord. 2011 Jan;44(1):81-90. doi: 10.1002/eat.20876. PMID 21080416